CLINICAL TRIAL: NCT02933463
Title: Clinical Effectiveness of Embrace Wetbond and Clinpro as Pits and Fissure Sealants in Young Permanent Molars, Randomized Clinical Trial
Brief Title: Clinical Effectiveness of Embrace Wetbond and Clinpro as Pits and Fissure Sealants in Young Permanent Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Abdullah agina, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Nagina
Record Dates: First submitted 2016-10-11; First posted 2016-10-14 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Caries
Keywords: children with high caries risk
MeSH Terms: interventions — Embrace WetBond; Clinpro Sealant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- embrace wetbond sealant (Experimental): moisture tolerant resin based, have same properties of other sealant
  Interventions: Other: Embrace Wetbond
- clinpro sealant (Active Comparator): is a dental resin, with low viscosity , fluoride releasing with a unique patented color change.
  Interventions: Other: Clinpro sealant

INTERVENTIONS:
Other: Embrace Wetbond — not require an additional bonding agent hydrophilic, fluoride releasing
  Arms: embrace wetbond sealant
Other: Clinpro sealant
  Arms: clinpro sealant

SUMMARY:
This study is designed to clinically evaluate the retention and development of caries when using self-priming (Embrace wetbond) and conventional flowable composite (Clinpro) as pit and fissure sealant in young first permanent molars.

DETAILED DESCRIPTION:
The aim of this study is designed to clinically evaluate the retention and development of caries when using self-priming (Embrace Wetbond) and conventional flowable composite (Clinpro) as pit and fissure sealant in young first permanent molars.

PICO:

P: children aged 6-9 years old with high caries risk.

I: Embrace Wetbond.

C: Clinpro seal.

O:

Primary outcome: Retention of sealant; Device of measurement: questionnaire; unit: binary.

Secondary outcome: Retention and development of caries; Device of measurement: Modified simonsen's criteria; Unit: scoring system (0-4) tactile and visual examination.

ELIGIBILITY:
Inclusion Criteria:

* children aged 6-9 years
* children with high caries risk
* cooperative children
* fully erupted first permanent molars

Exclusion Criteria:

* children with hypoplastic teeth
* partially erupted
* uncooperative children
* children with carious molars.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Retention of sealant | 6 months
  device for measurement: will make a questionnaire for the patients , unit of measurement: binary ( yes/no)

SECONDARY OUTCOMES:
Retention and development of caries | 6 months
  device of measurement: simonsen's criteria, unit of measurement: scoring system from 0-4 by tactile and visual examination.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Hamdy, professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aleksejuniene J, Brondani MA, Pattanaporn K, Brukiene V. Best practices for dental sealants in community service-learning. J Dent Educ. 2010 Sep;74(9):951-60. PMID 20837736
- [Background] Al-Jobair A. Scanning electron microscope analysis of sealant penetration and adaptation in contaminated fissures. J Indian Soc Pedod Prev Dent. 2013 Jul-Sep;31(3):169-74. doi: 10.4103/0970-4388.117970. PMID 24021327
- [Background] Bhat PK, Konde S, Raj SN, Kumar NC. Moisture-tolerant resin-based sealant: A boon. Contemp Clin Dent. 2013 Jul;4(3):343-8. doi: 10.4103/0976-237X.118394. PMID 24124301
- [Background] Bhatia MR, Patel AR, Shirol DD. Evaluation of two resin based fissure sealants: a comparative clinical study. J Indian Soc Pedod Prev Dent. 2012 Jul-Sep;30(3):227-30. doi: 10.4103/0970-4388.105015. PMID 23263426
- [Background] Deery C, Fyffe HE, Nugent ZJ, Nuttall NM, Pitts NB. General dental practitioners diagnostic and treatment decisions related to fissure sealed surfaces. J Dent. 2000 Jul;28(5):313-8. doi: 10.1016/s0300-5712(00)00004-x. PMID 10785296
- [Background] Kane B, Karren J, Garcia-Godoy C, Garcia-Godoy F. Sealant adaptation and penetration into occlusal fissures. Am J Dent. 2009 Apr;22(2):89-91. PMID 19626971
- [Background] Morales-Chavez MC, Nualart-Grollmus ZC. Retention of a resin-based sealant and a glass ionomer used as a fissure sealant in children with special needs. J Clin Exp Dent. 2014 Dec 1;6(5):e551-5. doi: 10.4317/jced.51688. eCollection 2014 Dec. PMID 25674325
- [Background] Rohr M, Makinson OF, Burrow MF. Pits and fissures: morphology. ASDC J Dent Child. 1991 Mar-Apr;58(2):97-103. PMID 2050885
- [Background] Reddy VR, Chowdhary N, Mukunda KS, Kiran NK, Kavyarani BS, Pradeep MC. Retention of resin-based filled and unfilled pit and fissure sealants: A comparative clinical study. Contemp Clin Dent. 2015 Mar;6(Suppl 1):S18-23. doi: 10.4103/0976-237X.152932. PMID 25821368
- [Background] Schlueter N, Klimek J, Ganss C. Efficacy of a moisture-tolerant material for fissure sealing: a prospective randomised clinical trial. Clin Oral Investig. 2013 Apr;17(3):711-6. doi: 10.1007/s00784-012-0740-2. Epub 2012 May 3. PMID 22552593
- [Background] Khatri SG, Samuel SR, Acharya S, Patil S, Madan K. Retention of Moisture-tolerant and Conventional Resin-based Sealant in Six- to Nine-year-old Children. Pediatr Dent. 2015 Jul-Aug;37(4):366-70. PMID 26314605
- [Background] Going RE, Loesche WJ, Grainger DA, Syed SA. The viability of microorganisms in carious lesions five years after covering with a fissure sealant. J Am Dent Assoc. 1978 Sep;97(3):455-62. doi: 10.14219/jada.archive.1978.0327. PMID 279600
- [Background] Mitchell DA, Mitchell L. Oxford Handbook of Clinical Dentistry (4th edition). New York: Oxford University Press; 2005.
- [Background] Ratnaditya A, Kumar MG , Jogenddrra SS,et al. Clinical evaluation of retention in hydrophobic and hydrophilic pit and fissure sealants-A Two Year Follow-Up Study. Journal of young pharmacist.2015;7(3):171.
- [Background] Strassler HE and O'Donnell JP. A unique moisture tolerant resin based pit and fissure sealant.2008.
- [Background] Pinkham J, Casamassimo P. Pediatric Dentistry. Infancy through Adolescence. 4 th ed. New Delhi: Saunders; 2005.
- [Background] Welburg R, Duggal H and Hosey M (Eds). Paediatric dentistry: treatment of dental caries in the preschool child. (3rd ed), 138-41.OXFORD UNIVERSITY PRESS, 2005.